CLINICAL TRIAL: NCT02377687
Title: Is Life Worth Living After Major Emergency GI Surgery? Patient Reported Outcome in Elderly Emergency Surgery Patients
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Line Toft Tengberg, MD, Hvidovre University Hospital
Other Study IDs: 2012-58-0004
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Emergency; Surgery
Keywords: Emergency surgery; HRQoL; Elderly
MeSH Terms: conditions — Emergencies | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly >75 years: all patients aged ≥ 75 having an emergency GI laparotomy or laparoscopy
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study

SUMMARY:
To study the impact of emergency high risk GI surgery on HRQOL in elderly patients, seventy-five years or above and to explore the patients' experience with the informed consent process and the status 6 months after surgery.

DETAILED DESCRIPTION:
We will identify all patients aged ≥ 75 having an emergency GI laparotomy or laparoscopy between the 1st of November 2014 and the 30st of April 2015.

The first part of the study will take place in the first postoperative week, while the patient is in hospital. After consent we will ask both patient and relatives/caregivers questions concerning the preoperative course and the informed consent. We will ask for permission to call the patients for a followup (the second part of the study) 5-7 months after discharge and permission to contact their closest relative. The closest relative is chosen by the patient and will after consent be asked the same questions in the first postoperative week and after 6 months.

The second part of the study will be initiated with a letter with SF-36 and an additional questionnaire . The SF-36 will be returned by letter. We will contact the patients by telephone 2 weeks after sending the letter ask them the questions from the additional questinaire.

We will compare the results from the SF-36 with age-matched controls (Data from the Danish SF-36 Manual).

If the patient is not capable of answering the questionnaires, the primary reason is noted (e.g. suffering from dementia or didn't speak Danish, dead).

We will aim at a 6 month follow-up period after discharge allowing a range from 5-7 months. Data acquisition will be done in the fall 2014 until late 2015.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 75 having an emergency GI laparotomy or laparoscopy between the 1st of November 2014 and the 30st of April 2015. We will also include reoperations after elective surgery (major bleeding, anastomotic leakage etc.) and endoscopic procedures converted during the intervention (upper GI-bleeding, unsuccessful stenting of obstructing colorectal cancer etc.).

Exclusion Criteria:

* appendectomies, negative laparoscopy/laparotomy, laparoscopic cholecystectomy, acute hernias without strangulation, sub-acute internal hernia after Roux-en-Y gastric bypass surgery, sub-acute IBD-surgery and sub-acute Colorectal Cancer-surgery. Sub-acute is defined as planned in less than 48 hours.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will identify all patients aged ≥ 75 having an emergency GI laparotomy or laparoscopy between the 1st of November 2014 and the 30st of April 2015. We will also include reoperations after elective surgery (major bleeding, anastomotic leakage etc.) and endoscopic procedures converted during the intervention (upper GI-bleeding, unsuccessful stenting of obstructing colorectal cancer etc.).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
HRQoL | 6 months after surgery

SECONDARY OUTCOMES:
Functional status | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bay-Nielsen, DMSc, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No